CLINICAL TRIAL: NCT02639442
Title: Clinical Study for the Evaluation of the Safety and Initial Performance of the ClearRing System for the Treatment of Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProArc Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA-CP-10
Record Dates: First submitted 2015-12-17; First posted 2015-12-24 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Benign ProstaticHyperplasia (BPH)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ClearRing™ (Experimental): subjects will undergo general/spinal/local block anesthesia and cystoscopy and/or x-ray evaluation. One to three implants will be transplanted into the patient prostate, followed by cystoscopy for results evaluation
  Interventions: Device: ClearRing™

INTERVENTIONS:
Device: ClearRing™

SUMMARY:
The ProArc Medical ClearRing™ system is a prostatic reshaping device that is designed to treat Lower Urinary Tract Symptoms (LUTS) due to BPH.

During the procedure an implant is delivered into the prostate tissue obstructing the urethra and restricting urine flow. The delivery system uses an electro-cutting blade to perform a circular and superficial incision, in which the implant is placed. Such an implant, with the shape of an open ring, expands the obstructed area, reducing the fluid obstruction through the prostatic urethra.

DETAILED DESCRIPTION:
The proposed study will be conducted on BPH patients, candidates for TURP and will aim to evaluate the ability of the ClearRing™ to improve BPH symptoms while conforming to safety of the procedure.

In the proposed study the implants will be inserted by a dedicated delivery system with the aid of resectoscope. Electrical current will be administered by off-the-shelf CE Mark diathermy that passes through the system to cut and pave the ring course.

The proper positioning of the implants will be evaluated by cystoscopy or TRUS and following implant positioning the device will be withdrawn.

The delivery tool, the implants, resectoscope and the diathermy equipment will be supplied by ProArc Ltd.

ELIGIBILITY:
Inclusion Criteria:

1. Male 50 years of age and up to 85 years old.
2. Diagnosed with symptomatic benign prostatic hyperplasia (BPH)
3. International Prostate Symptom Score (IPSS) >13
4. Peak flow rate ≤ 12 ml/sec (with voided volume ≥ 125ml)
5. Subject is in good general health.
6. Subject understands and has signed the study informed consent form.
7. PSA according to the American Urological Association) AUA) guideline.

Exclusion Criteria:

1. Subjects who are known to be infected with Hepatitis B, Hepatitis C, or HIV viruses.
2. Subject allergic to nickel or titanium
3. Concomitant participation in another study
4. Diagnosed with Cancer except of BCC or SCC of the skin
5. Any medical condition at the investigator discretion that may interfere with the procedure.
6. Patient with coagulopathy due to medications or congenital
7. Patient is taking steroids
8. Previous prostate surgery
9. Compromised renal function due to obstructive uropathy
10. Urinary Tract Infection (UTI)
11. Intravesical lobe (based on ultrasound and/or cystoscopy and/or medical history)
12. Prostate volume (based on Trans Rectal Ultrasound) > 80g
13. American Society of Anesthesiologists score (ASA)≥3
14. Known neurogenic bladder
15. Implanted electronic device such as pacemaker/CRT/ICD/DBS.
16. Recent myocardial infarction (less than three months)

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
The frequency and severity of all treatment-related adverse events | up to 3 months after procedure day

SECONDARY OUTCOMES:
Changes in Qmax | change from baseline until 3 months FU visit
  measured by Uroflowmetry
Changes in Post Void Residual | change from baseline until 3 months FU visit
  measured by Ultra-Sound
Changes in LUTS symptoms | change from baseline until 3 months FU visit
  evaluated by patient's questionnaires (IPSS)
Changes in LUTS symptoms | change from baseline until 3 months FU visit
  evaluated by patient's questionnaires ( BPHII)
Changes in LUTS symptoms | change from baseline until 3 months FU visit
  evaluated by patient's questionnaires ( IIEF)

OTHER OUTCOMES:
Duration of Catheter use post procedure | until 12 months post procedure
Long term safety evaluation | until 12 months post procedure
  AE collection

CONTACTS AND LOCATIONS:
Locations (2):
- Rambam MC, Haifa, Israel
- Department of Urology, Pauls Stradins Clinical University Hospital, Riga, Latvia

IPD SHARING:
Plan to Share IPD: Undecided